CLINICAL TRIAL: NCT00751920
Title: Comparative Evaluation of MRI and MDCT for the Detection of Metastic Pulmonary Nodules
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The sponsor-investigator relocated to a different institution and was not able to continue the study.
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000010635
Record Dates: First submitted 2008-09-10; First posted 2008-09-12 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Metastatic Pulmonary Nodules
Keywords: Magnetic Resonance Imaging; Pediatrics; Multi-Detector Computed Tomography; Computed Tomography; Detection
MeSH Terms: conditions — Multiple Pulmonary Nodules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: Enhanced MRI Scan

INTERVENTIONS:
Procedure: Enhanced MRI Scan — Following the detection of a pulmonary nodule(s) with the unenhanced MRI scan, the subjects will then be injected with the contrast agent, Magnevist, and have a dynamic enhanced MRI scan of the largest pulmonary nodule.

SUMMARY:
The purpose of this study is to apply the techniques of dynamic MRI imaging enhancement to research participants with one or more pulmonary nodule to determine if meaningful information about the nature of the nodule can be obtained. This data will then be compared with follow up information about nodule growth or histology obtained by biopsy or surgical resection.

DETAILED DESCRIPTION:
The gold standard for investigating the detection of pulmonary metastases is Multi-Detector Computed Tomography (MDCT). Computed Tomography (CT) is routinely used in the staging of pediatric patients with primary tumors which commonly metastasize to the lungs (with approximate percentage incidence of pulmonary metastases at presentation) are Ewing's sarcoma (15-20%), osteosarcoma (15-20%), Wilm's Tumor (10%), rhabdomyosarcoma (10%), and hepatoblastoma (10%). However, CT scanning has two central limitations. Firstly, it carries associated radiation risks. This risk is increased if multiple scans need to be performed during treatment and follow up. This is of particular concern in children who frequently have curable disease and may have years to live with the radiation risk. Secondly, CT is limited in its ability to distinguish between benign and malignant nodules.

Recently, Magnetic Resonance Imaging (MRI) of the lung has been shown to be a feasible alternative to CT for the detection of pulmonary metastases in adults with sensitivities and specificities of over 90% for the detection of nodules 5mm or larger. It has also shown promise in the characterization of nodules as benign or malignant. Since MRI does not involve radiation, it may prove to be a preferable imaging technique for children. We wish to evaluate the potential for MRI to complement or even replace CT in the imaging of pulmonary metastatic disease in children.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 2-18 years of age
* Patients who present themselves to the Department of Diagnostic Imaging at the Hospital for Sick Children for CT of the thorax
* Patients undergoing a CT of the thorax for detection of lung metastases following diagnosis of a solid tumor or suspected solid tumor
* Patients who present themselves for initial diagnosis or at follow up CT for progression
* Able to give informed consent (parents or patients)

Exclusion Criteria:

* Usual exclusion criteria for MRI (e.g. pacemaker, ocular metal, claustrophobia)
* Have any known allergy to one or more of the ingredients in the study contrast agents; have a history of hypersensitivity to any metals or chelates of gadolinium; have a history of allergies or bronchial asthma; use beta blockers, have cardiovascular disease; or have anaphylactic reactions
* Have moderate-to-severe renal impairment (defined as having a GFR/ eGFR < 60 mL/min)
* Have sickle cell anemia
* MRI of the chest requiring sedation or general anesthesia
* Known pregnancy or breast feeding
* Renal failure
* Patient uncooperative during a MRI without sedation or anesthesia (unless already receiving this for MRI of another body region)
* Children under the age of 2 will not be eligible for intravenous contrast

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2008-08; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
MRI sensitivity for the detection of pulmonary nodule(s) greater than 3mm in size (diameter) compared to CT | One hour

SECONDARY OUTCOMES:
How accurate MRI is at distinguishing between benign and malignant pulmonary nodules. | One hour

CONTACTS AND LOCATIONS:
Overall Officials: Paul Babyn, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada